CLINICAL TRIAL: NCT00791869
Title: Pharmacogenetics of Bupropion Metabolism
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: H133-31868; U01DA020830 (NIH)
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Metabolism; Pharmacokinetics
Keywords: bupropion; smoking; pharmacokinetics; Pharmacokinetics of bupropion
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the investigators research is to see if variants in a particular gene (named CYP2B6) affect how the body metabolizes (breaks down) certain medications, including the drug bupropion. Bupropion is widely used in the treatment of depression and for helping people quit smoking. Genes are portions of DNA that code for particular proteins in the body. The investigators are studying the gene that codes for a protein called CYP2B6. Differences in the structure of the gene are called variants and may mean that a person metabolizes a drug faster or slower than a person with a different variant.

DETAILED DESCRIPTION:
Bupropion is widely used in the treatment of depression and for smoking cessation. It's most abundant metabolite, hydroxybupropion, may be responsible for most of the therapeutic effect of bupropion under conditions of long term dosing. Because the primary enzyme involved in metabolism of bupropion to hydroxybupropion is the liver enzyme CYP2B6, we propose to study the effect of different CYP2B6 genotypes on the metabolism of bupropion. These data will guide the use of genotypes as a surrogate for measuring drug blood levels in studying genetic determinants of outcomes for bupropion treatment.

A minimum of Forty-four subjects with 4 different CYP2B6 genotypes will participate in a 7-day study in which they take bupropion as outpatients for 6 days (to achieve steady state drug levels) and then come to the San Francisco General Hospital (SFGH) Clinical Research Center for a 1-day admission during which multiple blood and urine samples will be collected for pharmacokinetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 65 years
* Gender: Either
* Ethnic/Racial Group: Any
* Smoking Status: Both smokers and non-smokers are eligible
* CYP2B6 genotype: CYP2B6 *1/*1 (11 subjects); *4, *5 and *6 alleles (11 each) [44 subjects total] Up to 15 additional subjects may be studied with genotypes that do not fall into one of the primary groups.

Exclusion Criteria:

* Medical: Exclude most any chronic illness requiring regular medication.
* Cardiac: History of angina or other serious heart disease; ECG abnormalities on screening.
* Hypertension: screening visit BP of 150/95 or more after 5 min rest
* Respiratory: Asthma - acceptable if in remission, otherwise exclude.
* Systemic: "Morbidly Obese" Exclude if BMI > 35
* Diabetes: By history
* Chronic Active Hepatitis: By history; elevated Liver Function Tests
* Cancers: By history
* Pregnancy/breastfeeding: By history; positive urine pregnancy test
* Seizures: individuals with a history of seizures will be excluded (risk factor for bupropion-induced seizures)
* Eating Disorders: individuals with a history of eating disorders will be excluded (risk factor for bupropion-induced seizures)
* Head Trauma: individuals with a history of head trauma will be excluded (risk factor for bupropion-induced seizures)
* Other tobacco users (pipe, cigar, chewing tobacco, snuff users
* Medications/Supplements: General Exclusion = "any regular oral and/or prescription drug use"; current use of oral contraceptives or other female hormones.
* Drug/alcohol use: no alcohol abuse by history, no regular recreational drug use, any intravenous drug abuse, recent history of Treatment program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects with selected CYP2B6 genotypes.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2008-06; Primary Completion 2010-03 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) for bupropion | 0, 4, 8, 12, 16,24 hours from steady state
  Subjects took bupropion daily for 7 days as outpatients prior to the study day to allow them to reach steady state concentrations of bupropion and its metabolites. The time frame shown is measured from 08:00 on the morning of inpatient admission.

CONTACTS AND LOCATIONS:
Overall Officials: Neal L Benowitz, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital-Clinical Research Ward, San Francisco, California, United States